CLINICAL TRIAL: NCT04075253
Title: Acute Effect of One Single Bout of High Intensity Exercise. A Substudy of the Study on Physical Activity and Ventricular Arrhythmias
Brief Title: Acute Effect of One Single Bout of High Intensity Exercise on the Tendency for Ventricular Arrhythmia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1592-b
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Tachycardia, Ventricular; Defibrillators, Implantable
Keywords: Exercise Training
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VO2 peak test (Experimental): All participants enrolled in the planned study on physical activity and ventricular arrhythmias and on baseline will complete an exercise treadmill test to determine VO2 peak
  Interventions: Behavioral: VO2 peak testing

INTERVENTIONS:
Behavioral: VO2 peak testing — Exercise on treadmill starts with ~4km/h at 0% inclination before inclination is increased to 4% and speed kept unchanged. Inclination will then be increased with two percent approximately after each minute until exhaustion.
  Other Names: Cardiopulmonary Exercise Testing (CPET)

SUMMARY:
This study will evaluate the acute effect of one single bout of high intensity exercise on the tendency for ventricular arrhythmia.

DETAILED DESCRIPTION:
This study is a substudy of a planned study involving participants with an implantable cardioverter defibrillator (ICD), who will be randomly assigned to either take part in a exercise program for 12 weeks or serve as control and live as usual (Clinical Trials Unique Protocol ID: 2018/1592). In that study all participants will complete an exercise treadmill test to determine maximum oxygen uptake (VO2 peak).

In this study we wish to examine the acute effect of one single bout of high intensity exercise (i.e the VO2 peak test) on the tendency for ventricular arrhythmia. The study will evaluate changes in ICD-parameters and the number of premature ventricular contractions the first 24 hours after VO2 peak testing compared to the average number of the 48 hours prior to the test.

The study will also examine if the acute effect after VO2 peak testing alters after completing 12 weeks of aerobic interval training or control respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ICD and dilated cardiomyopathy or coronary heart disease as cause for implantation
* ICD implanted at St Olavs hospital, Trondheim

In case of difficulties with patient inclusion for the study, the criteria might be broadened to include patients with idiopathic ventricular arrhythmia as cause for implantation.

Exclusion Criteria:

* inability to accomplish the exercise program due to serious comorbidity or to participate in regular training within the next 3 months due to other reasons
* signs of severe cardiac ischemia or persistent ventricular tachycardia during individualized treadmill O2 peak test, which after individual assessment is to be found at risk
* comorbidity where endurance training at more than moderate intensity is discouraged
* severe cardiac valve disease
* planned surgery within the next 3 months
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Tendency for ventricular arrhythmia | 24 hours
  Measured by changes in the number of premature ventricular contractions the first 24 hours after VO2 peak testing compared to the average number of the 48 hours prior to the test. Registered on a 72 hours Holter monitoring

SECONDARY OUTCOMES:
Changes in ICD-parameters during a single bout of high intensity exercise (VO2 peak test) | 24 hours
  Evaluated by changes in number of inappropriate shocks
Changes in ICD-parameters during a single bout of high intensity exercise (VO2 peak test) | 24 hours
  Evaluated by changes in stimulation threshold
Changes in ICD-parameters during a single bout of high intensity exercise (VO2 peak test) | 24 hours
  Evaluated by changes in lead impedance
Changes in ICD-parameters during a single bout of high intensity exercise (VO2 peak test) | 24 hours
  Evaluated by changes in atrial and ventricular refractory period
Changes in ICD-parameters during a single bout of high intensity exercise (VO2 peak test) | 24 hours
  Evaluated by changes in restitution time of the sinus node
Changes in ICD-parameters during a single bout of high intensity exercise (VO2 peak test) | 24 hours
  Evaluated by changes in refractory period of the AV-node
Changes in acute effect of one single bout of high intensity exercise on tendency for ventricular arrhythmia after either 3 months of interval exercise or control | Baseline and after 12 weeks
  Measured by changes in the number of premature ventricular contractions the first 24 hours after VO2 peak testing compared to the average number of the 48 hours prior to the test. Registered on a 72 hours Holter monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Rune Wiseth, MD, Prof, Study Director — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for all primary and secondary outcome measures will be made available after deidentiﬁcation and publication
Time Frame: After publication
Access Criteria: Not yet decided